CLINICAL TRIAL: NCT05859815
Title: The Role of Mechanical Diagnosis and Therapy in the Classification and Management of Concussion
Brief Title: The Role of Mechanical Diagnosis and Therapy in the Management of Concussion
Status: Recruiting | Type: Observational
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Michael Brown, Clinical Assistant Professor, State University of New York at Buffalo
Other Study IDs: STUDY00006666
Record Dates: First submitted 2023-03-22; First posted 2023-05-16 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Brain Concussion; Mild Traumatic Brain Injury
Keywords: Mechanical Diagnosis and Therapy; Directional Preference; Repeated Movements
MeSH Terms: conditions — Brain Concussion | interventions — Physical Therapy Modalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Directional preference responder: This group is comprised of participants who responded to repeated movements in a direction (e.g., neck flexion) that significantly improved their symptoms and/or their ability to move their head/neck.
  Interventions: Behavioral: Physical Therapy
- Directional preference non-responder: This group is comprised of participants who did not respond to repeated movements in any specific direction that significantly improved their symptoms and/or their ability to move their head/neck.
  Interventions: Behavioral: Physical Therapy

INTERVENTIONS:
Behavioral: Physical Therapy — As part of their normal care, participants will receive any combination of the following interventions to address their specific needs identified during the initial evaluation: cervical spine repeated movements (active range of motion), cervical spine stabilization exercise, aerobic exercise, motor control training, oculomotor/vestibular rehabilitation, stretching, soft-tissue mobilization, joint mobilization, and postural re-education activities.

SUMMARY:
The purpose of this study is to examine the role of a Mechanical Diagnosis and Therapy (MDT) examination in identifying participants diagnosed with concussion who display a directional preference compared to who don't display a directional preference.

DETAILED DESCRIPTION:
Directional preference describes the clinical phenomenon where a specific direction of repeated movement and / or sustained position results in a clinically relevant improvement in symptoms. This improvement is usually accompanied by an improvement in function or mechanics or both. Its presence and relevance is determined over 2-3 visits. This study aims to identify the proportion of participants with concussion who present with a directional preference during the course of physical therapy. A secondary aim of this study is to investigate whether directional preference is associated with the eventual patient related outcomes following care.

ELIGIBILITY:
Inclusion Criteria:

* Age = 13 - 65
* Complaints of neck pain, headache, or dizziness associated with a diagnosis of concussion or mild TBI
* Ability to read/write English
* Referral from physician

Exclusion Criteria:

* Age less than 13 or greater than 65
* Cause of symptoms is result of a work-related accident or motor vehicle accident
* Receiving concurrent treatment from a chiropractor or massage therapist
* Glasgow Coma Scale less than 12
* Lesion on head CT/MRI
* Focal neurological deficits associated with serious spinal pathology (fracture, infection, tumor, vertebrobasilar insufficiency)
* Inability to or unwilling to exercise as part of usual PT care
* Unable to read/write English
* History of osteopenia/osteoporosis or cancer

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of patients who have been diagnosed with a concussion and referred for outpatient physical therapy services.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-07-20 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Directional preference classification | Through study completion, up to 1 year.
  Outcome represents the patient's directional preference at the time of discharge from care. Patients will be classified as directional preference responders or non-responders.

SECONDARY OUTCOMES:
Post-Concussion Symptom Scale | Through study completion, up to 1 year.
  The PCSS is a patient self-reported outcome measure that measures the amount of interference associated with a concussion across four domains: physical, cognitive, emotion, and sleep. The measure consists of 22 questions that relate to post-concussive symptoms. The measure uses a 7-point Likert scale, where 0 = no symptoms and 6 = severe symptoms. The greatest possible score is 132 and the lowest score is 0. Higher scores indicate higher severity of post-concussive symptoms.
Neck Disability Index | Through study completion, up to 1 year.
  The NDI is a patient self-reported outcome measure that measures the amounts of pain interference and self-reported disability related to neck pain. The measure consists of ten questions in the following domains: pain intensity, personal care, lifting, reading, sleeping, work, recreation, reading, concentration, and headaches. Each item is rated on a 0 to 5 scale, where 0 = no disability and 5 = complete disability. The highest possible raw score equals 50 points, the lowest possible score equals 0. The raw scores can also be converted to a percentage from 0 to 100%. Higher scores indicate higher levels of self-reported disability.
Dizziness Handicap Inventory | Through study completion, up to 1 year.
  The DHI is a patient self-reported outcome measure that measures the impact of dizziness on daily life. The DHI consists of 25 items measuring the impact of dizziness across three domains: functional (9 questions,= 36 points), emotional (9 questions = 36 points), and physical (7 questions = 28 points). Each item is rated on a 3 point scale (yes = 4, sometimes = 2, no = 0). Item scores are summed, with a possible total of 100 points. The best possible score is a 0. Higher scores indicate greater perceived handicap due to dizziness.

OTHER OUTCOMES:
Return to sport/activity | Up to 1 year
  This outcome represents the number of days it takes a patient to return to their prior level of participation in sport/activity
Number of treatments | Up to 1 year
  This outcome represents the number of physical therapy visits they completed before being discharged by the physician or physical therapist.

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Brown, DPT, PhD, Principal Investigator — University at Buffalo
Locations (2):
- United States (2):
  - Goodlife Physical Therapy, Orland Park, Illinois
  - Summit Healthplex Physcial Therapy/Niagara Falls Memorial Medical Center, Niagara Falls, New York

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers.